CLINICAL TRIAL: NCT02794584
Title: Precision Assessment of Perioperative Effectiveness and Safety of Transthoracic Minimally Invasive Hybrid Closure for Pediatric Ventricular Septal Defects
Brief Title: Hybrid Closure of Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHD-Nanjing
Record Dates: First submitted 2016-05-25; First posted 2016-06-09 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pediatric Ventricular Septal Defects
MeSH Terms: interventions — Sufentanil; Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Off-pump hybrid closure (Active Comparator): Hybrid closure is that a periventricular technique uses an occluding device to closure ventricular septal defects of patients through the delivery system by transthoracic minimally invasive small incision without cardiopulmonary bypass.
  Interventions: Drug: sufentanil anesthesia; Procedure: Hybrid closure
- Control (Placebo Comparator): Control group: Conventional closure of ventricular septal defects was aided with cardiopulmonary bypass.
  Interventions: Drug: sufentanil anesthesia; Procedure: Control

INTERVENTIONS:
Drug: sufentanil anesthesia — Anaesthesia is maintained by inhaled isoflurane in concentrations 0.7-0.8 % end-tidal with additional sufentanil injected during surgery, as required. During extracorporal circulation patients receive isoflurane via a vaporizer incorporated in the extracorporeal gas supply in the same concentrations.
  Other Names: Sufentanil, Sufenta, (R-30730)
Procedure: Hybrid closure — Hybrid closure of ventricular septal defects through the delivery system without cardiopulmonary bypass by transthoracic minimally invasive small incision.
  Other Names: TTMI: Transthoracic Minimally Invasive
  Arms: Off-pump hybrid closure
Procedure: Control — Surgical closure of ventricular septal defects with cardiopulmonary bypass by routine open thoracotomy.
  Other Names: CPB: cardiopulmonary bypass
  Arms: Control

SUMMARY:
Ventricular septal defect (VSD) is one of the most common pediatric congenital malformations. In recent years, in view of the rapid rise of transthoracic minimally invasive hybrid closure for pediatric VSD in the clinical practice, precision assessment of perioperative its effectiveness and safety has already become an important issue that must be solved. On the basis of echocardiography, integrating with characteristics associated critical care, the investigators focus on precision assessment of perioperative effectiveness and safety of transthoracic hybrid closure for pediatric VSD, compared with conventional surgical sternotomy repair with cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of perimembranous ventricular septal defect, muscular ventricular septal defect, doubly committed subarterial VSD by transesophageal echocardiogram (TEE) with VSD size 5-12mm;
* no significant aortic insufficiency or aortic valve prolapse.

Exclusion Criteria:

* confirmed pulmonary hypertension (systolic pulmonary arterial pressure >75mmHg or pulmonary vascular resistance >8.0 Wood U/m2);
* more than mild degree of aortic regurgitation and obvious aortic valve prolapse;
* preoperative congestive heart failure;
* other coexisting cardiac anomalies;
* infective endocarditis.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Myocardial injury as measured by cardiac troponin I serum | 7 days postoperatively after cardiac surgery
Respiratory dysfunction as measured by PaO2 | 7 days postoperatively after cardiac surgery

SECONDARY OUTCOMES:
All cause mortality | 7 days postoperatively after cardiac surgery

OTHER OUTCOMES:
Number of participants with right bundle branch block assessed by ECG | 7 days postoperatively after cardiac surgery
Left ventricular ejection fractions | 7 days postoperatively after cardiac surgery
Extravascular lung water index | 7 days postoperatively after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hai-tao Gu, MD, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

REFERENCES:
- [Background] Amin Z, Danford DA, Lof J, Duncan KF, Froemming S. Intraoperative device closure of perimembranous ventricular septal defects without cardiopulmonary bypass: preliminary results with the perventricular technique. J Thorac Cardiovasc Surg. 2004 Jan;127(1):234-41. doi: 10.1016/j.jtcvs.2003.08.023. PMID 14752435
- [Derived] Liu H, Lu FX, Zhou J, Yan F, Qian SC, Li XY, Zheng SQ, Chen JQ, Zhong JS, Feng QL, Ding T, Fan J, Gu HT, Liu XC. Minimally invasive perventricular versus open surgical ventricular septal defect closure in infants and children: a randomised clinical trial. Heart. 2018 Dec;104(24):2035-2043. doi: 10.1136/heartjnl-2017-312793. Epub 2018 Jun 25. PMID 29941505